CLINICAL TRIAL: NCT06971354
Title: Tratamiento de la rumiación: Estudio Aleatorizado, Paralelo y Controlado
Brief Title: Treatment of Rumination
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)057-2025
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Rumination Syndrome
MeSH Terms: conditions — Rumination Syndrome | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental): Three biofeedback sessions will be administered during the first three weeks of the intervention period. In each session, participants will receive a standardized meal and undergo training to control abdominal and thoracic muscular activity. This training will be guided by a trained operator using original audiovisual materials and hands-on techniques. Regurgitation episodes will be recorded by participants using an event marker. Following each session, participants will be instructed to perform the same exercises before and after breakfast, lunch, and dinner throughout the four-week intervention period.
  Interventions: Behavioral: Biofeedback
- Placebo (Placebo Comparator): Three treatment sessions will be conducted during the first three weeks of the intervention period. In each session, participants will receive a placebo capsule prior to a standardized meal and will be instructed to record the number of regurgitation episodes using an event marker. Following each session, participants will be asked to take a placebo capsule before each meal throughout the four-week intervention period.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Behavioral: Biofeedback — Three sessions of biofeedback before and after a standardized meal.
  Arms: Biofeedback
Dietary Supplement: Placebo — Three sessions of placebo followed by standardized meal.
  Arms: Placebo

SUMMARY:
Background: Rumination syndrome is characterized by the involuntary regurgitation of previously ingested food from the stomach to the mouth, triggered by an unintentional contraction of the abdominal muscles along with simultaneous relaxation of the esophageal sphincters. Based on this mechanism, a biofeedback technique targeting muscular activity has been developed and shown to be effective. However, such techniques are often complex and not widely accessible.

Hypothesis: Rumination can be effectively treated using a simplified, non-instrumental biofeedback technique based on cognitive intervention.

Objective: To evaluate the effectiveness of a non-instrumental biofeedback technique incorporating cognitive intervention for the treatment of rumination. The methodology will build on prior studies, employing a more streamlined biofeedback approach.

Methods: Participants will be assigned to parallel groups with balanced sex distribution. The study will compare responses to biofeedback versus a control intervention. Over a four-week period, each participant will undergo three treatment sessions:

The biofeedback group will be trained to control abdominothoracic musculature through cognitive intervention, supported by original visual materials, both before and after a standardized test meal.

The control group will receive a placebo capsule prior to the test meal, and regurgitation episodes will be recorded.

Following the initial session, biofeedback participants will continue with daily exercises, while control participants will take a placebo with each meal. Treatment response will be assessed by comparing outcomes before and after the intervention. After post-treatment assessment, control group participants will be offered the opportunity to receive biofeedback therapy.

Relevance: This project aims to determine the efficacy of a simplified mechanistic intervention for rumination. If successful, this approach could be adopted in additional healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Rumination syndrome

Exclusion Criteria:

* Relevant organic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of rumination events after a challenge meal measured by an event marker. | 4 weeks
  Each regurgitation event will be registered by the patient using an event marker.

SECONDARY OUTCOMES:
Number of self perceived rumination events | 4 weeks
  Number of rumination events measured by questionnaires administered daily for 7 days before and at the end of treatment.
Number of rumination events | 1 month
  Number of rumination events measured by questionnaires administered daily for 7 days, 1 month after treatment.
Number of rumination events | 3 months
  Number of rumination events measured by questionnaires administered daily for 7 days, 3 months after treatment.
Number of rumination events | 6 months
  Number of rumination events measured by questionnaires administered daily for 7 days, 6 months after treatment.
Quantity of meal regurgitated | 4 weeks
  The quantity of the standardized meal that is regurgitated will be recorded, and the proportion of regurgitated to ingested meal will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Serra, M.D., Principal Investigator — Vall d'Hebron Research Institute, Barcelona, 08035
Locations (1):
- Vall d'Hebron Research Institute, Barcelona, Spain